CLINICAL TRIAL: NCT06826885
Title: The Safety and Efficacy of IMPT or IMRT for Breast Cancer: A Prospective Observational Study
Brief Title: Safety and Efficacy of IMPT or IMRT for Breast Cancer
Acronym: SEPPT-BC
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Collaborators: Shandong Cancer Hospital and Institute (Other); Sichuan Cancer Hospital and Research Institute (Other); Cancer Hospital Chinese Academy of Medical Science, Shenzhen Center (Other); Tongji Hospital (Other)
Responsible Party: Principal Investigator, JIAYI CHEN, Chair of Radiation Oncology Department, Ruijin Hospital
Other Study IDs: RJBC- SEPPT-BC
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-12

CONDITIONS: Breast Cancer; Proton Therapy; Intensity Modulated Radiation Therapy; Efficacy and Safety; Radiotherapy, Adjuvant
Keywords: postoperative radiotherapy; preoperative radiotherapy; IMPT; IMRT; breast cancer; efficacy; toxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Arm1: Postoperative radiotherapy: Patients who indicated postoperative radiotherapy using IMRT or IMPT.
  Interventions: Radiation: Postoperative radiotherapy
- Arm2：Preoperative radiotherapy: Patients who indicated preoperative radiotherapy using IMRT or IMPT.
  Interventions: Radiation: Preoperative Radiotherapy
- Arm3：Definitive radiotherapy: Patients who indicated definitive radiotherapy using IMRT or IMPT.
  Interventions: Radiation: Definitive Radiotherapy

INTERVENTIONS:
Radiation: Postoperative radiotherapy — Radiotherapy was administered using IMPT or IMRT. The target volume includes the ipsilateral whole breast, chest wall, and/or regional lymph nodes. A hypofractionated regimen of 40-42.5 Gy (RBE) in 15-16 fractions is preferred. A conventional fractionated regimen of 45-50.4 Gy (RBE) at 1.8-2 Gy per fraction in 25-28 fractions or an ultra-hypofractionated regimen of 26 Gy (RBE) in 5 fractions is also allowed. A tumor bed boost will be provided to patients with high-risk factors following breast-conserving surgery, at the discretion of the radiation oncologist. The tumor bed boost regimen may consist of a sequential boost of 10-16 Gy (RBE) in 5-8 fractions, or 10-13.35 Gy (RBE) in 4-5 fractions or 10.4 Gy (RBE) in 2 fractions, or a simultaneous integrated boost of 48-49.5 Gy (RBE) in 15-16 fractions.
  Groups: Arm1: Postoperative radiotherapy
Radiation: Preoperative Radiotherapy — Radiotherapy was administered using IMPT or IMRT. The target volume includes the ipsilateral whole breast, chest wall, and/or regional lymph nodes. A hypofractionated regimen of 40-42.5 Gy (RBE) in 15-16 fractions is preferred. A conventional fractionated regimen of 45-50.4 Gy (RBE) at 1.8-2 Gy per fraction in 25-28 fractions or an ultra-hypofractionated regimen of 26 Gy (RBE) in 5 fractions is also allowed.
  Groups: Arm2：Preoperative radiotherapy
Radiation: Definitive Radiotherapy — Radiotherapy was delivered using IMPT or IMRT. The target volume encompassed the ipsilateral whole breast and regional lymph nodes. A hypofractionated regimen of 40-42.5 Gy (RBE) in 15-16 fractions was preferred. Alternatively, a conventional fractionated regimen of 45-50.4 Gy (RBE) at 1.8-2 Gy per fraction in 25-28 fractions or an ultra-hypofractionated regimen of 26 Gy (RBE) in 5 fractions was permitted. Dose escalation was applied in high-risk areas, resulting in a total prescribed dose exceeding 66 Gy (RBE) when calculated as equivalent doses in 2-Gy fractions (EQD2), with an α/β ratio of 4.
  Groups: Arm3：Definitive radiotherapy

SUMMARY:
The purpose of this trial is to compare the toxicities and efficacy of intensity-modulated proton therapy (IMPT) and intensity-modulated radiation therapy (IMRT) for breast cancer patients indicated for radiotherapy including preoperative radiotherapy, postoperative radiotherapy, or definitive radiotherapy. IMPT or IMRT will be administered to the whole breast, chest wall, and/or regional lymph nodes. A boost dose will be delivered in patients with high-risk area, at the discretion of the radiation oncologist. Eligible breast cancer patients will be followed for at least 5 years to assess acute and late radiation induced toxicities, loco-regional recurrence, overall survival, distant metastasis, and quality of life.

DETAILED DESCRIPTION:
Eligible breast cancer patients will receive either preoperative, postoperative, or definitive radiotherapy based on the MDT's recommendation. Patients with indications for treatment will receive either the IMPT or IMRT technique. The specific technique will be chosen based on the benefits of IMPT, patient preference, and reimbursement policies after discussion between the doctor and the patient. The primary endpoint is the occurrence of any acute radiation-induced toxicities of grade ≥2. Patients will be monitored for at least five years to evaluate acute and late radiation-induced toxicities, loco-regional recurrence, overall survival, distant metastasis, and quality of life.

ELIGIBILITY:
Inclusion Criteria

* Aged ≥18 years old
* Karnofsky Performance Status (KPS) score ≥70
* Histologically confirmed breast cancer with indications for preoperative radiotherapy, postoperative radiotherapy, or definitive radiotherapy as determined by the treating physician.
* ER (estrogen-receptor), PR (progesterone-receptor), HER2 (human epidermal growth factor receptor 2), and Ki67 testing must be performed on the primary breast tumor.
* Women of child-bearing potential must agree to use adequate contraception starting 1 month before study treatment and throughout the duration of study participation.
* Ability to understand and willingness to participate in the research and sign the informed consent form.

Exclusion Criteria

* Pregnant or lactating women.
* Severe non-neoplastic medical comorbidities that may interfere with treatment or study participation.
* Active collagen vascular disease or other autoimmune disorders that could significantly increase the risk of radiation toxicity.
* Patients with contraindications to undergoing IMPT or IMRT, such as severe claustrophobia that cannot be managed or inability to remain immobilized during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients aged ≥18 years with histologically confirmed disease and indications for preoperative radiotherapy, postoperative radiotherapy, or definitive radiotherapy, as determined by the treating physician, who are willing to receive radiotherapy using IMPT or IMRT.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Complication Rate of ≥Grade 2 Acute Radiation-Induced Toxicity | 6 months
  Acute radiation-induced toxicities will be assessed and recorded from the start of radiotherapy to six months after its completion. Evaluations will occur weekly during treatment, and at 2 weeks, 4 weeks, 3 months, and 6 months post-treatment. The assessment will utilize the Radiation Therapy Oncology Group (RTOG)/European Organization for Research and Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring Schema and the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Complication Rate of ≥Grade 2 Late Radiation-induced Toxicity | 5 years
  From six months after the completion of radiotherapy to five years post-treatment, any late radiation-induced toxicity will be assessed and recorded every six months during the first two years, and annually thereafter. Assessments will utilize the Radiation Therapy Oncology Group (RTOG) /European Organization for Research on Treatment of Cancer (EORTC) Late Radiation Morbidity Scoring Schema and CTCAE 5.0
Locoregional recurrence | 5 years
  Any first recurrence confirmed by histology or cytology within the ipsilateral breast or chest wall and/or regional nodes area (including supraclavicular, infraclavicular, axillary, or internal mammary lymph nodes)
Distant Metastasis-Free Survival (DMFS) | 5 years
  The duration from the date of enrollment to the occurrence of any breast tumor recurrence at distant sites, death from any cause, or the last follow-up.
Invasive Recurrence-Free Survival (iRFS) | 5 years
  The duration from the date of enrollment to the occurrence of the first invasive breast tumor recurrence, death from any cause, or the last follow-up.
Overall Survival (OS) | 5 years
  The duration from the date of enrollment to the date of death from any cause or the last follow-up.
Pathologic Complete Response (pCR) Rate After Preoperative Radiotherapy | 8-12 weeks
  The percentage of patients who achieve ypT0/is and ypN0 (no invasive residual in the breast or lymph nodes) after preoperative radiotherapy.
Progression-Free Survival (PFS) After Definitive Radiotherapy | 5 years
  The duration from the initiation of definitive radiotherapy to the earliest occurrence of any of the following events:
  Disease Progression: As determined by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
  Death: From any cause. Last Follow-Up: If neither progression nor death occurs during the study period.
Objective Response Rate (ORR) After Definitive Radiotherapy | 3 to 12 months
  The percentage of patients who achieve a complete response (CR) or partial response (PR) to definitive radiotherapy, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Disease Control Rate (DCR) After Definitive Radiotherapy | 3 to 12 months
  The percentage of patients who achieve a complete response (CR), partial response (PR), or stable disease (SD) to definitive radiotherapy, as assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.

OTHER OUTCOMES:
Quality of Life using self-administered questionnaire EORTC QLQ-C30 | 5 years
  The time from the date of enrollment to 5 years after completion of radiotherapy, Quality of life will be assessed before radiotherapy, every 6 months during the first 2 years and annually thereafter using self-administered questionnaire EORTC QLQ-C30
Number of Participants with Excellent or Good Cosmetic Outcomes Following Breast-Conserving Surgery | 5 years
  The duration from the date of enrollment to five years after the completion of radiotherapy will be assessed for cosmetic outcomes. Evaluations will occur before radiotherapy, every 6 months during the first two years, and annually thereafter. Cosmetic outcomes will be assessed using the Allegheny General Modification of the Harvard/National Surgical Adjuvant Breast and Bowel Project (NSABP)/RTOG scoring scale, which classifies patients into the following four categories:
  Excellent: Minimal or no difference in size or shape of the treated breast compared to the untreated breast.
  Good: Slight difference in size or shape of the treated breast. Fair: Obvious difference in size or shape of the treated breast. Poor: Marked change in size or shape of the treated breast.
Patient-Reported Outcomes (PRO) survey | 5 years
  PRO are measures that capture patients' perceptions of their health status, symptoms, and quality of life directly from the patients, without interpretation by healthcare providers. In this study, PROs will be assessed at baseline before the initiation of radiotherapy, then every 6 months during the first 2 years, and annually thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Cai, MD, Principal Investigator — Ruijin Hospital; Jia-Yi Chen, PhD, MD, Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided